CLINICAL TRIAL: NCT02608476
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of Cortexolone 17α-Propionate (CB-03-01) Cream, 1% Applied Twice Daily for 12 Weeks in Subjects With Facial Acne Vulgaris
Brief Title: A Study to Evaluate the Safety and Efficacy of CB-03-01 Cream, 1% in Subjects With Facial Acne Vulgaris (26)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-03-01/26
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: acne; clascoterone; anti-androgen
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB-03-01 cream (Experimental): CB-03-01 cream, 1% applied twice daily for 12 weeks
  Interventions: Drug: CB-03-01 cream, 1%
- Vehicle cream (Placebo Comparator): Vehicle cream applied twice daily for 12 weeks
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: CB-03-01 cream, 1% — CB-03-01 (cortexolone 17α-propionate) is a steroidal antiandrogen that is being developed as a 1% cream for the topical treatment of acne vulgaris.
  Other Names: cortexolone 17α-propionate; clascoterone (USAN, INN)
  Arms: CB-03-01 cream
Drug: Vehicle cream — Vehicle cream manufactured to mimic look and feel of CB-03-01 but without the active ingredient cortexolone 17α-propionate.
  Arms: Vehicle cream

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of CB-03-01 cream, 1%, versus the vehicle cream applied twice daily for 12 weeks in subjects with facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female, 9 years of age or older. Females must be post-menopausal, surgically sterile, or using highly effective birth control methods. Women of child-bearing potential must have a negative urine pregnancy test (UPT) at the Screening/Baseline Visit.
2. Subject has provided written and verbal informed consent/assent. A subject under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing.
3. Subject has an Investigator's Global Assessment (IGA) score of 3 (moderate) or 4 (severe) [0 (clear) to 4 (severe) scale].
4. Subject has facial acne vulgaris with at least 30 to a maximum of 75 inflammatory lesions (papules, pustules, and nodules) and 30 to a maximum of 100 non-inflammatory lesions (open and closed comedones).
5. Subject and parent/guardian (if applicable) are willing to comply with study instructions and return to the clinic for required visits.
6. Subject has used the same type and brand of make-up, other facial products (exclusive of RX/OTC acne cleansers) and hair products (e.g., shampoo, gel, hair spray, mousse, etc.) for at least one (1) month prior to the Baseline Visit and agrees to continue his/her other general skin and hair care products and regimen for the entire study.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical or systemic therapy.
3. Subject has greater than two (2) facial nodules.
4. Subject has nodulocystic acne.
5. Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. Subject is currently enrolled in an investigational drug or device study.
7. Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (Baseline).
8. Subject has facial hair that could interfere with the study assessments in the opinion of the investigator.
9. Subject and parent/guardian (if applicable) are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
10. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
11. Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
12. Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.
13. Subject has used any of the prohibited topical anti-acne treatments or procedures prior to the study unless appropriate washout period is documented.
14. Subject has used used any of the prohibited systemic anti-acne medications prior to the study unless appropriate washout period is documented.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Cassiopea, Study Director — Cassiopea S.p.A.
Locations (52):
- United States (12):
  - Clear dermatology & Aesthetic Center, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Belleair Research Center, Pinellas Park, Florida
  - Arlington Dermatology, Arlington Heights, Illinois
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - Sadick Research Group, LLC, New York, New York
  - Skin Specialty Dermatology, New York, New York
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
- Bulgaria (8):
  - Site 3521, Plovdiv
  - Site 3523, Sofia
  - Site 3525, Sofia
  - 3520, Sofia
  - Site 3524, Sofia
  - Site 3519, Sofia
  - Site 3526, Sofia
  - Site 3522, Varna
- Georgia (6):
  - Site 9923, Batumi
  - Site 9924, Kutaisi
  - Site 9921, Tbilisi
  - Site 9920, Tbilisi
  - Site 9922, Tbilisi
  - Site 9925, Zugdidi
- Poland (13):
  - 4819, Bydgoszcz
  - Site 4814, Częstochowa
  - Site 4822, Częstochowa
  - 4815, Katowice
  - Site 4811, Katowice
  - Site 4821, Krakow
  - Site 4815, Krakow
  - Site 4813, Krakow
  - Site 4820, Lodz
  - Site 4823, Osielsko
  - Site 4816, Rzeszów
  - Site 4812, Szczecin
  - Site 4818, Warsaw
- Romania (10):
  - Site 4033, Sector 2, Bucharest
  - Site 4034, Sector 2, Bucharest
  - Site 4031, Sector 3, Bucharest
  - Site 4029, Sector 6, Bucharest
  - Site 4028, Târgovişte, Jud. Dambovita
  - Site 4036, Bucharest
  - Site 4035, Bucharest
  - Site 4032, Craiova
  - Site 4037, Iași
  - Site 4030, Sibiu
- Serbia (3):
  - Site 8138, Belgrade
  - Site 8137, Belgrade
  - Site 8136, Novi Sad

REFERENCES:
- [Derived] Hebert A, Eichenfield L, Thiboutot D, Stein Gold L, Vassileva S, Mihaylova Y, Cartwright M, Moro L, Fragasso E, Han J, Squittieri N, Mazzetti A. Efficacy and Safety of 1% Clascoterone Cream in Patients Aged > 12 Years With Acne Vulgaris. J Drugs Dermatol. 2023 Feb 1;22(2):174-181. doi: 10.36849/JDD.7000. PMID 36745367
- [Derived] Piszczatoski CR, Powell J. Topical Clascoterone: The First Novel Agent for Acne Vulgaris in 40 Years. Clin Ther. 2021 Oct;43(10):1638-1644. doi: 10.1016/j.clinthera.2021.08.007. Epub 2021 Oct 2. PMID 34607697
- [Derived] Hebert A, Thiboutot D, Stein Gold L, Cartwright M, Gerloni M, Fragasso E, Mazzetti A. Efficacy and Safety of Topical Clascoterone Cream, 1%, for Treatment in Patients With Facial Acne: Two Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2020 Jun 1;156(6):621-630. doi: 10.1001/jamadermatol.2020.0465. PMID 32320027

RESULTS

PARTICIPANT FLOW:
Groups:
- CB-03-01 Cream: CB-03-01 cream, 1% applied twice daily for 12 weeks
  Cortexolone 17α-propionate (USAN/INN: clascoterone) is a steroidal antiandrogen that is being developed as a
  1% cream for the topical treatment of acne vulgaris.
Period: Overall Study
Arm/Group | CB-03-01 Cream | Vehicle Cream
Started | 369 | 363
Completed | 302 | 282
Not Completed | 67 | 81
Not completed — Withdrawal by Subject | 30 | 37
Not completed — Lost to Follow-up | 24 | 24
Not completed — Adverse Event | 2 | 8
Not completed — Withdrawal by Parent/Guardian | 5 | 4
Not completed — Noncompliance with treatment | 1 | 5
Not completed — Lack of Efficacy | 3 | 1
Not completed — Other | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population; defined as all subjects randomized and whom received at least one dose of study medication, including vehicle.
Groups:
- Total: Total of all reporting groups
Arm/Group | CB-03-01 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 369 | 363 | 732
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.3 (5.6) | 19.0 (5.4) | 19.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243 | 221 | 464
  Male | 126 | 142 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 9 | 29
  Not Hispanic or Latino | 349 | 354 | 703
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 6 | 13
  White | 357 | 348 | 705
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 2 | 6
Baseline IGA [Count of Participants; unit: Participants] — Investigator's Global Assessment (IGA)
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 305 | 313 | 618
    4 - Severe | 64 | 50 | 114
Baseline Acne Lesion Counts [Mean (Standard Deviation); unit: lesions]
  Non-inflammatory lesions | 62.8 (21.4) | 63.3 (20.5) | 63.1 (21.0)
  Inflammatory lesions | 42.9 (12.2) | 41.3 (11.0) | 42.1 (11.6)
  Total Lesions | 105.7 (25.8) | 104.6 (24.2) | 105.2 (25.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Success in Investigator's Global Assessment (IGA)
Description: Percentage of subjects in each treatment group achieving "success" at Week 12, with "success" defined as an IGA score of "clear (score=0)" or "almost clear (score=1)" and at least a two-point reduction in IGA compared to Baseline.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population, which included all randomized subjects
Measure: Number; unit: Percentage of subjects
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
Percentage of subjects | 20.3 | 6.5

2. Primary Outcome: Change From Baseline in Non-inflammatory Lesion (NIL) Counts
Description: Absolute change from Baseline in non-inflammatory lesion counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: Non-inflammatory lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
Non-inflammatory lesions | -19.4 [-22.1 to -16.7] | -10.8 [-13.6 to -8.0]

3. Primary Outcome: Change From Baseline in Inflammatory Lesion (IL) Counts
Description: Absolute change from Baseline in inflammatory lesion counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: Inflammatory lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
Inflammatory lesions | -20.0 [-21.7 to -18.3] | -12.6 [-14.3 to -10.8]

4. Secondary Outcome: Change From Baseline in Total Lesion Counts
Description: Absolute change from Baseline in total lesions counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: total lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
total lesions | -40.0 [-43.8 to -36.2] | -23.6 [-27.8 to -19.5]

5. Secondary Outcome: Percent Change From Baseline in Total Lesion Counts
Description: Percent change from Baseline in total lesions counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
percent change | -37.3 [-41.1 to -33.6] | -22.1 [-26.1 to -18.1]

6. Secondary Outcome: Percent Change From Baseline in Non-inflammatory Lesion Counts
Description: Percent change from Baseline in non-inflammatory lesions count in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
percent change | -29.3 [-33.7 to -24.9] | -15.6 [-20.3 to -10.9]

7. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts
Description: Percent change from Baseline in inflammatory lesions count in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 369 | 363
percent change | -46.9 [-50.9 to -42.8] | -29.6 [-33.9 to -25.3]

8. Other Pre Specified Outcome: Local Site Reactions
Description: Local Site Reactions (LSRs) including telangiectasia, skin atrophy, striae rubrae, erythema, edema, scaling/dryness, stinging/burning, and pruritus scored by frequency and severity at every visit (Baseline, Weeks 4, 8, and 12).
Time Frame: Baseline, Weeks 4, 8, and 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from screening visit, Baseline (Day 1) and up to Week 12/early termination.
Description: The Safety population was used for all analyses which comprised of all participants enrolled in the study and applied at least on dose of the test article.
Arm/Group | CB-03-01 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/369 | 0/363
Serious Adverse Events (participants affected / at risk) | 0/369 | 1/363
Other Adverse Events (participants affected / at risk) | 21/369 | 34/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream (N=369) | Vehicle Cream (N=363)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream (N=369) | Vehicle Cream (N=363)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02608476/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT02608476/SAP_001.pdf